CLINICAL TRIAL: NCT01650129
Title: An Open-labelled, Randomised, Parallel Group, Multicentre, Safety and Efficacy Study of NN-X14Mix50 (BIAsp50) in a Twice Daily Regimen in Type 2 Diabetic Subjects
Brief Title: Safety and Efficacy of Biphasic Insulin Aspart 50 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1352
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp (Experimental)
  Interventions: Drug: biphasic insulin aspart 50
- BHI (Experimental)
  Interventions: Drug: biphasic human insulin 50

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — Administered subcutaneously (s.c., under the skin) twice daily for 24 weeks. Injected immediately before breakfast and dinner
  Arms: BIAsp
Drug: biphasic human insulin 50 — Administered subcutaneously (s.c., under the skin) twice daily for 24 weeks. Injected 30 minutes before breakfast and dinner
  Arms: BHI

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the safety and efficacy of biphasic insulin aspart (BIAsp) 50 (NN-X14Mix50) compared with biphasic human insulin (BHI) 50 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Subjects with insulin treated for at least 24 weeks
* HbA1c maximum 11.0%
* Body mass index (BMI) below 30.0 kg/m^2
* Patients who have the skill of self-injection of insulin, and are able and willing to perform self-monitoring blood glucose (SMBG) and are able to take measures against hypoglycaemic episodes

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Subjects with proliferative retinopathy or preproliferative retinopathy diagnosed within the last 12 weeks, or receiving photocoagulation therapy within the last one year
* Impaired hepatic function
* Impaired renal function
* Cardiac diseases
* Uncontrolled hypertension
* Subjects with history of severe allergic or severe hypersensitive reactions
* Total daily insulin dose at least 100 IU
* Treatment with oral hypoglycaemic agentsvwithin the last 4 weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2000-12-13 (Actual); Primary Completion 2001-10-18 (Actual); Study Completion 2001-10-18 (Actual)

PRIMARY OUTCOMES:
Glycosylated haemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Occurrence of adverse event(s)
Blood glucose
Incidence of hypoglycaemic episodes
Change from baseline in insulin antibodies
Insulin doses

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com